CLINICAL TRIAL: NCT03403335
Title: Mindfulness Practices for Healthcare Professional Trainees
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: American Psychological Association (APA) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: HM20012397
Record Dates: First submitted 2018-01-11; First posted 2018-01-18 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-05

CONDITIONS: Stress
MeSH Terms: interventions — Health Personnel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Based Practices for Health Care Professionals (Experimental)
  Interventions: Behavioral: Mindfulness Based Practices for Health Care Professionals in Training
- Control Group (No Intervention)

INTERVENTIONS:
Behavioral: Mindfulness Based Practices for Health Care Professionals in Training — Eight weekly sessions including didactic lecture, discussion, homework, gentle yoga, and meditation and mindfulness exercises
  Arms: Mindfulness Based Practices for Health Care Professionals

SUMMARY:
A newly developed intervention, Mindfulness Based Practices for Health Care Professionals in Training: Clinical Applications, will be piloted to determine the feasibility and accessibility within this population. The purpose of the proposed study is to assess the change in perceived stress at work/school and psychological symptomology; i.e., depression, stress, emotion regulation, and dispositional mindfulness, from pre to post intervention in health care professional students and when compared to a matched control group.

DETAILED DESCRIPTION:
The proposed study aims to investigate an 8-week intervention: Mindfulness Based Practices for Health Care Professionals in Training: Clinical Applications. During the intervention, participants will engage in didactic education, experiential mindfulness practices, including gentle yoga, and group dialogue. The aim of the study is to investigate the feasibility of this intervention in producing measurable differences between the participants and matched controls on their perception of their well-being and clinical work.

ELIGIBILITY:
Inclusion Criteria:

* Students/faculty from any health care department at VCU

Exclusion Criteria:

* Anyone who is not a student/faculty from a health care department at VCU

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2018-02-09 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-04-28 (Actual)

PRIMARY OUTCOMES:
Change in burnout | administered at baseline, post-intervention (8 weeks), and 3 month post-intervention follow-up
  Assessed using Maslach Burnout Inventory a 22 item screening tool with higher values indicating more burnout
Change in depressive symptoms | administered at baseline, post-intervention (8 weeks), and 3 month post-intervention follow-up
  Assessed using Patient Health Questionnaire 9. 9-items with lower values indicating less depression
Change in state anxiety | administered at baseline, post-intervention (8 weeks), and 3 month post-intervention follow-up
  Assessed using State Trait Anxiety Inventory -- a 20 item measure with some items reverse scored and higher scored indicating higher state anxiety
Change in ruminative thinking | administered at baseline, post-intervention (8 weeks), and 3 month post-intervention follow-up
  Assessed using Rumination Response Scale -- a 10 item measure with higher scores indicating higher rumination
Change in stress | administered at baseline, post-intervention (8 weeks), and 3 month post-intervention follow-up
  Assessed using Perceived Stress Scale -- a 14-item scale with higher scores indicating higher levels of stress
Change in dispositional mindfulness | administered at baseline, post-intervention (8 weeks), and 3 month post-intervention follow-up
  Assessed using Five Facet Mindfulness Questionnaire -- a 39-item measure of 5 domains of mindfulness in daily life, with higher scores indicating higher levels of mindfulness
Change in cognitive functioning | administered at baseline and post-intervention (8 weeks)
  Assessed using Trail Making Test A & B -- a brief task requiring respondents to connect numbered dots and then switch between number and letters, speed and accuracy are both recorded

SECONDARY OUTCOMES:
Change in interprofessional attitudes measure | administered at baseline, post-intervention (8 weeks), and 3 month post-intervention follow-up
  Assessed using Interprofessional Team Training Assessment -- a 22-item measure and Student Perceptions of Physician-Pharmacist Interprofessional Clinical Education -- a 10-item measure; both with higher scores indicating more positive attitudes toward interprofessional training
Follow-up Interview of Perceptions of Mindfulness and Interprofessional Education | assessed at 3-month post-intervention follow-up
  qualitative interview and exploration -- participants will spend approximately 30 minute by phone being interviewed on their experiences with the intervention especially in the context of healthcare and interprofessional education

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Rybarczyk, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

REFERENCES:
- [Derived] Braun SE, Mladen SN, Luberto CM, Kinser PA. Maintenance of Effects and Correlates of Changes Following Mindfulness for Interdisciplinary Health Care Professional Students. Integr Med Rep. 2022 Sep 1;1(1):177-185. doi: 10.1089/imr.2021.0012. Epub 2022 Sep 7. PMID 36212225